CLINICAL TRIAL: NCT05386381
Title: Long Term Survivorship of Decompression Alone Versus Decompression With Fusion in Patients With Degenerative Lumbar Spondylolisthesis and Lumbar Canal Stenosis
Brief Title: Survivorship of Decompression Alone Vs Decomp With Fusion in DLS and LCS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1854
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Lumbar Spondylolisthesis Involving L4-L5
Keywords: Degenerative Lumbar Spondylolisthesis; Lumbar Canal Stenosis; Fusion; Decompression; Fenestration; Spinous Process Osteotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decompression alone: Patients undergone decompression surgery alone
- Decompression with fusion: Patient undergone decompression and lumbar fusion surgery

SUMMARY:
There has been a long-standing controversy on the operative treatment of Degenerative Lumbar Spondylolisthesis (DLS) with Lumbar Canal Stenosis (LCS), especially whether the addition of fusion to decompression is necessary. Many believe that decompression alone (D) by either using midline preserving fenestration techniques (fenestration by laminotomy and medial facetectomy) or with a spinous process osteotomy (SPO) is enough for treatment of patients with DLS while others believe that a fusion (D+F) should be added in all cases.

The study aims to determine if decompression alone performs better or worse in the long term than decompression with fusion in a large cohort of patients who have DLS with LCS. It also aims to determine if the decompression technique of midline-sparing fenestration or spinous process osteotomy make a difference to survival in cases of DLS with LCS.

DETAILED DESCRIPTION:
The study aims to utilize already obtained data from the clinical service, obtainable from the electronic patient records (EPR). It would be a retrospective review of data on patients with DLS treated operatively.

All data collected will be anonymized prior to any analysis. The primary outcome to be analyzed is the time to repeat surgery/procedure at the previously operated vertebral level. This will be regarded as failure of the original surgery and will be used in the survival analysis. All analysis will be done at the RJAH site. As the study will use anonymized data collected through the clinical service, individual patient consent will not be obtained.

All data used in this study has been obtained during the patients' routine clinical care and follow up. No further tests or scans other than routine patient care will be performed. The data for this study will be collected and anonymized before any statistics is performed. Only data for patients with DLS + LCS treated operatively between 1st January 2002 and 31st December 2006 that have had at least 15 years of follow up will be extracted. The data is currently stored on the Trust secure patient record system. As all the data will be anonymized no consents will be required. Data collected will include age, gender, date of admission, consultant, primary procedure date, length of hospital stay, date of death, type of surgery (fenestration/fenestration+fusion/spinous process osteotomy), fusion/no fusion, type of fusion (instrumented/non-instrumented/interbody), unilateral/bilateral, laminectomy/no laminectomy, number of levels, discectomy, post op complications, revision surgery, date of revision, coexisting problems.

Analysis of the data will address the following: Does difference in technique of lumbar decompression or adding fusion affect long term survivorship in degenerative lumbar spondylolisthesis with canal stenosis (DLS +LCS)? Does decompression alone perform better or worse in the long term than decompression with fusion in a large cohort of patients who have DLS with LCS. Does decompression technique of midline-sparing fenestration or spinous process osteotomy make a difference to survival in cases of DLS with LCS

Statistics The primary outcome which is the time to failure will be used to generate the Kaplan-Meier survival function for each of the three surgical techniques. The survival curves will then be compared using the Mantel-Cox (Log rank) test for statistical significance. Statistical significance will be set at p < 0.05. A sub group analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients with degenerative lumbar spondylolisthesis

Exclusion Criteria:

* Patients with spondylolysis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with degenerative lumbar spondylolisthesis treated operatively between 1st January 2002 and 31st December 2006 at Robert Jones and Agnes Hunt Orthopaedic Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to Revision | 15 years
  Duration between initial surgery and revision surgery at same level

CONTACTS AND LOCATIONS:
Overall Officials: olakunle J Alonge, MBBS, FWACS, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS FT
Locations (1):
- Robert Jones and Agnes Hunt Orthopedic Hospital, Oswestry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data only